CLINICAL TRIAL: NCT00006643
Title: Use of Single Photon Emission Computed Tomography (SPECT) as a Noninvasive Alternative to Liver Biopsies in Assessing Liver Involvement in Subjects Coinfected With HIV and Hepatitis C Virus (HCV)
Brief Title: Comparing Single Photon Emission Computed Tomography (SPECT) and Liver Biopsy to Evaluate the Liver in Patients With HIV and Hepatitis C Virus
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: ACTG A5096; AACTG A5096
Record Dates: First submitted 2000-12-06; First posted 2001-08-31 (Estimated); Last update posted 2008-07-30 (Estimated); Status verified 2003-06

CONDITIONS: HIV Infections; Hepatitis C
Keywords: Liver; Hepatitis C; Biopsy; Tomography, Emission-Computed, Single-Photon
MeSH Terms: conditions — HIV Infections; Hepatitis C

SUMMARY:
The purpose of this study is to find if the Single Photon Emission Computed Tomography (SPECT) scan is as effective as a liver biopsy (using a special needle to remove tissue from the liver) in examining liver damage in patients with HIV and hepatitis C virus (HCV).

A standard way to examine the liver for disease has been to perform a liver biopsy. The SPECT scan, which takes a picture of the liver, has been found to be effective in determining liver damage but studies need to be done in patients with hepatitis. This study will compare the effectiveness of the liver biopsy and SPECT scan in determining liver disease in patients with HIV and HCV. The SPECT scan might be a good replacement for the liver biopsy if it is found to be as good as or better than liver biopsies.

DETAILED DESCRIPTION:
Assessment with a liver biopsy is currently the standard of practice to determine the status of liver involvement in patients with HCV. A direct comparison between SPECT results and liver pathology has been examined in patients with liver disease other than infectious hepatitis. SPECT has been found to be more accurate than standard liver-spleen scans in assessing liver pathology. While current data suggest that liver pathology may correlate with SPECT, which specific SPECT parameters are predictive of certain hepatic pathology is unknown. The pilot study will compare SPECT parameters with the results of liver biopsies to determine the limitations of SPECT.

All screened patients are registered into Step 1, in which they receive a radioactive tracer injection and SPECT scan. Specific SPECT parameters will be measured to determine a grading scale corresponding to that used in liver biopsy results. Some patients undergoing a second liver biopsy in A5071 are enrolled into Step 2, with permission from protocol co-chairs, in which a pregnancy test and second SPECT scan are performed. Patients are reimbursed for completing each SPECT scan. SPECT scans or copies are reviewed to establish which parameters correspond to category E of the Knodell stage based on severity of fibrosis.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are enrolled in, or will soon enroll in, A5071. Patients may be eligible for the study if they are screening for A5071 and have a liver biopsy and SPECT scan but do not enter A5071. Patients who have stopped taking A5071 study drugs may also be eligible.
* Have had a liver biopsy, or will soon have a liver biopsy.
* Have a SPECT scan either before the liver biopsy or 2 weeks to 8 weeks after a liver biopsy.
* Intend to have the SPECT scan within 7 days of study entry.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are allergic to chemicals in the radioactive tracer used for the SPECT scan.
* Are pregnant or breast-feeding.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Shiramizu, Study Chair; Dickens Theodore, Study Chair
Locations (11):
- United States (11):
  - Stanford Univ Med Ctr, Stanford, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Hawaii, Honolulu, Hawaii
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Community Health Network Inc, Rochester, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ of Cincinnati, Cincinnati, Ohio
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Univ of Texas, Southwestern Med Ctr of Dallas, Dallas, Texas
  - Univ of Washington, Seattle, Washington